CLINICAL TRIAL: NCT01392001
Title: Evaluation of Glucocorticoid Sparing Effect in Patients Receiving RoActemra® for Rheumatoid Arthritis in Real Life.
Brief Title: An Observational Study of Glucocorticoid Use in Patients With Rheumatoid Arthritis on Treatment With RoActemra/Actemra (Tocilizumab)
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML25634
Record Dates: First submitted 2011-07-08; First posted 2011-07-12 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Cohort

SUMMARY:
This observational study will evaluate the glucocorticoid sparing effect after 12 months of treatment with RoActemra/Actemra (tocilizumab) in patients with rheumatoid arthritis. Data will be collected for 12 months after the initiation of treatment with RoActemra/Actemra from patients who had been on treatment with >5 mg prednisone or equivalent for at least 3 months .

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >/= 18 years of age
* Patients with rheumatoid arthritis for whom the rheumatologist decided to introduce RoActemra
* Patients taking more than 5 mg/day of oral prednisone (or equivalent) for at least 3 months

Exclusion Criteria:

* Participation in a clinical trial in rheumatoid arthritis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Rheumatoid arthritis patients on treatment with RoActemra/Actemra and > 5 mg/day prednisone (or equivalent)
Sampling Method: Probability Sample
Enrollment: 322 (Actual)
Dates: Start 2011-03; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Percentage of patients receiving </= 5 mg/day prednisone (or equivalent) after 12 months of treatment with RoActemra/Actemra | approximately 29 months

SECONDARY OUTCOMES:
Efficacy: Disease activity score (DAS 28) | approximately 29 months
Co-medications: dosage and treatment schedules | approximately 29 months
Patient reported outcome: European League against Rheumatism - Rheumatoid Arthritis Impact of Disease score (EULAR-RAID)/Health Assessment Questionnaire - Disease Index (HAQ-DI) | approximately 29 months
Safety: Incidence of adverse events | approximately 29 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (97):
- France (97):
  - Abbeville
  - Agen
  - Aix-en-Provence
  - Aix-les-Bains
  - Alençon
  - Amiens
  - Angers
  - Argenteuil
  - Auch
  - Aulnay-sous-Bois
  - Avignon
  - Bayonne
  - Belfort
  - Belley
  - Berck
  - Besançon
  - Blois
  - Bobigny
  - Bois-Colombes
  - Bondy
  - Bordeaux
  - Brest
  - Caen
  - Cahors
  - Cambrai
  - Cannes
  - Carcassonne
  - Chambray-lès-Tours
  - Clermont-Ferrand
  - Compiègne
  - Corbeil-essones
  - Corbeil-Essonnes
  - Dijon
  - Dole
  - Druex
  - Évian-les-Bains
  - Évreux
  - Évry
  - Fréjus
  - Gap
  - Gleizé
  - La Roche-sur-Yon
  - Laon
  - Lavaur
  - Le Coudray
  - Le Kremlin-Bicêtre
  - Libourne
  - Liévin
  - Lille
  - Limoges
  - Lomme
  - Lorient
  - Lyon
  - Maisons-Laffitte
  - Mandelieu-la-Napoule
  - Marseille
  - Meaux
  - Metz-Tessy
  - Montauban
  - Montpellier
  - Morlaix
  - Moulins
  - Mulhouse
  - Nanterre
  - Nantes
  - Narbonne
  - Nice
  - Niort
  - Nîmes
  - Paris
  - Perpignan
  - Pierre-Bénite
  - Poissy
  - Pontoise
  - Reims
  - Rodez
  - Roubaix
  - Saint-Chamond
  - Saint-Flour
  - Saint-Mandé
  - Saint-Nazaire
  - Saint-Priest-en-Jarez
  - Saint-Quentin
  - Salon-de-Provence
  - Ste Maxime
  - Suresnes
  - Thionville
  - Toulon
  - Toulouse
  - Tourcoing
  - Valenciennes
  - Vandœuvre-lès-Nancy
  - Vannes
  - Vienne
  - Villefranche-sur-Saône
  - Villeurbanne
  - Vlleneuve Sur Lot